CLINICAL TRIAL: NCT01002001
Title: Prospective Study to Evaluate Sleep Disturbance in Patients With Liver Disease Pre and Post Liver Transplantation
Brief Title: Sleep Disorders Pre and Post Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Health Network, Toronto (Other)
Responsible Party: George Therapondos, University Health Network,
Other Study IDs: REB 09-0459
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sleep disturbance and sexual dysfunction are common complaints of patients with cirrhosis . The term sleep disturbance describes insomnia, poor quality sleep, circadian rhythm disorders and obstructive sleep apnea and is associated with reduced health-related quality of life (HRQoL) score indices. Sleep and sexual disorders have only been formally evaluated in small studies in these patients and to date, no studies have objectively assessed these patients. In addition, no studies have been performed in these patients after liver transplantation. The investigators' hypothesis is that sleep and sexual disturbance is commonly seen in patients with advanced cirrhosis and improves after liver transplantation. However, despite this, HRQoL remain impaired because of residual sleep disturbance.This study will be unique in providing cross-sectional follow-up of patients with cirrhosis at baseline and after liver transplantation (> 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Comprehend and read English
* On liver transplantation list or post-liver transplantation

Exclusion Criteria:

* Non-English speaking
* < 18 years and > 85 yrs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the pre and post-transplantation liver clinics
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Sleep disturbances in patients with advanced cirrhosis | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: George Therapondos, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada